CLINICAL TRIAL: NCT04459156
Title: Fiber Metabolism in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Director, Texas A&M University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2019-0832
Record Dates: First submitted 2020-06-22; First posted 2020-07-07 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Aging
Keywords: fiber metabolism; short chain fatty acid production rates
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Participants (Experimental): healthy control subjects
  Interventions: Dietary Supplement: Fiber Inulin; Dietary Supplement: Placebo Maltodextrin
- Chronic Obstructive Pulmonary Disease patients (Experimental): Established diagnosis of Chronic Obstructive Pulmonary Disease
  Interventions: Dietary Supplement: Fiber Inulin; Dietary Supplement: Placebo Maltodextrin
- Healthy Young Participants (Experimental): healthy young subjects with age 18-30 years old
  Interventions: Dietary Supplement: Fiber Inulin; Dietary Supplement: Placebo Maltodextrin

INTERVENTIONS:
Dietary Supplement: Fiber Inulin — Commercially available inulin is provided as powder. The following doses will be administered twice daily (with breakfast and dinner): Day 1-2: 5-g; Day 3: 7.5-g; Day 4: 10-g; Day 5: 12.5-g; Day 6-7: 15-g. All supplements are commercially available.
Dietary Supplement: Placebo Maltodextrin — Commercially available maltodextrin is provided as powder. The following doses will be administered twice daily (with breakfast and dinner): Day 1-2: 5-g; Day 3: 7.5-g; Day 4: 10-g; Day 5: 12.5-g; Day 6-7: 15-g. All supplements are commercially available.

SUMMARY:
The impact of fiber intake on short chain fatty acid (SCFA) metabolism has not been studied in subjects suffering from COPD. The purpose of this study is to compare changes in SCFA metabolism after inulin vs. placebo intake in COPD patients to healthy matched controls. This protocol is an extension of a recent study about whole-body SCFA production rates in COPD patients. The investigators hypothesize that a short-term fiber supplementation increases SCFA production in COPD patients.

DETAILED DESCRIPTION:
Dietary fibers are indigestible carbohydrates, which are present in several daily foods such as beans, legumes, whole grain products, and whole fruits and vegetables. The Food and Drug Administration recommends a daily fiber uptake of 25 g. However, in 2009-2010 the mean fiber intake of US adults was 17 g/day. Fiber cannot be digested by human enzymes and reach the colon undigested. Depending on the chemical structure (solubility, degree of polymerization) of the fiber, it can or cannot be fermented by the intestinal bacteria. Insoluble, unfermented fibers such as cellulose help to prevent constipation by enhancing bowel movement and the transit time of the feces. Most soluble fibers like inulin can be fermented by intestinal bacteria. During the bacterial fermentation short-chain fatty acids (SCFA) such as acetate (C2), propionate (C3), and butyrate (C4) are produced. The production is highest in the proximal colon where the abundance of fiber is the highest. The colonocytes absorb more than 90 % of the SCFAs, the rest is excreted with the feces. Most of the butyrate is oxidized in the colonocytes, being their main energy source. Propionate gets metabolized by the liver. In particular acetate enters the systemic circulation and might have anti-inflammatory and immune modulating effects. Indole and isovalerate are products of bacterial amino acid fermentation. Indole is solely produced by bacterial enzymes from the essential amino acid tryptophan (TRP) and isovalerate from branched-chain amino acids.

In COPD an enhanced pulmonary inflammatory response causes a combination of small airways disease (e.g., obstructive bronchiolitis) and/or a destruction of lung parenchyma (emphysema). This leads to a progressive and persistent airflow limitation. It has been shown that a healthy overall diet as well as a diet high in fiber can be associated with a good lung function and a decreased COPD prevalence. A diet rich in fermentable fiber altered the gut and lung microbiota composition in mice, mainly through a decrease in the Firmicutes-to-Bacteroidetes-ratio, which was accompanied by elevated concentrations of circulating SCFAs. These mice were protected against allergic inflammation in the lungs. Previous human research has demonstrated that the composition of the intestinal microbiota influences the asthma risk and it was associated with early life exacerbations in cystic fibrosis, which demonstrates a gut-lung cross-talk. Halnes et al. found a significantly reduced airway inflammation in asthma patients four hours after the ingestion of a meal containing soluble fiber and prebiotics compared to a placebo meal. Stable tracer studies are needed to examine the colonic production and metabolic fate of SCFAs in healthy and ill subjects.

The intestinal microbiota of older individuals is less diverse, has a higher interindividual variability, and lower SCFA production capacity compared to younger adults. Hence, a dysbiosis of the intestinal microbiota could be involved in the development of several age-related chronic systemic diseases, such as sarcopenia and lower muscle quality or cognitive dysfunction. These age-related impairments are associated with a reduced physical performance and elevated risk for falls, fractures, physical disability and mortality. Dysbiosis of the intestinal microbiota (i.e. an altered microbial composition and function) might contribute to the development of sarcopenia by modulating muscle size, composition, and function. Moreover, SCFAs, metabolites produced by beneficial bacteria, help maintaining cognitive function and psychological well-being through their anti-inflammatory and gene regulating properties. Hence, nutritional interventions, such as fiber supplementation, must be studies as a modulator of microbial composition and SCFA production rate, as well as the subsequent effects on muscle and cognitive health and overall well-being.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female according to the investigator's or appointed staff's judgment
* Ability to walk, sit down and stand up independently
* Age 45 - 100 years for healthy control subjects
* Age 18 - 30 years for healthy, young adults
* Ability to lay in supine or elevated position for 1.5 hours
* No diagnosis of COPD
* Willingness and ability to comply with the protocol

Inclusion criteria COPD subjects:

* Ability to walk, sit down and stand up independently
* Age 45 - 100 years
* Ability to lie in supine or elevated position for 1.5 hours
* Diagnosis of moderate to very severe chronic airflow limitation and compliant to the following criteria: FEV1 < 70% of reference FEV1
* Clinically stable condition and not suffering from a respiratory tract infection or exacerbation of their disease (defined as a combination of increased cough, sputum purulence, shortness of breath, systemic symptoms such as fever, and a decrease in FEV1 > 10% compared with values when clinically stable in the preceding year) at least 4 weeks prior to the first test day
* Shortness of breath on exertion
* Willingness and ability to comply with the protocol

Exclusion criteria all subjects:

* Any condition that may interfere with the definition 'healthy subject' according to the investigator's judgment (healthy subjects only)
* Insulin dependent diabetes mellitus
* Established diagnosis of malignancy
* History of untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Presence of fever within the last 3 days
* Use of short course of oral corticosteroids within 4 weeks preceding study day
* Dietary or lifestyle characteristics:

  * Daily use of fiber supplements 1 week prior to the first test day
  * Daily use of protein supplements 5 days prior to each test day
* Indications related to interaction with study products:

  * Known allergy to inulin or inulin products
  * Known hypersensitivity to inulin or maltodextrin or any of its ingredients
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* (Possible) pregnancy
* Already enrolled in another clinical trial and that clinical trial interferes with participating in this study
* Any other condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Whole body short-chain fatty acid production rates by plasma samples | Weeks 1, 2, 4, and 5
  Differences and changes in whole body SCFA production rates in COPD patients and healthy older and young adults after administration of stable-isotope labeled short-chain fatty acids.
Intestinal microbiota composition by stool sample collection using Shallow Shotgun Sequencing | Collection up to 24 hours before study visits of weeks 1, 2, 4, and 5
  Differences and changes in intestinal microbiota composition in COPD patients and healthy older and young adults using Shallow Shotgun Sequencing

SECONDARY OUTCOMES:
Intestinal integrity markers by stool samples | Weeks 1, 2, 4, and 5
  Differences and changes in fecal zonulin levels in COPD patients and healthy older and young adults.
Exhalation of CO2 from short-chain fatty acid oxidation | Weeks 1, 2, 4, and 5
  Differences and changes in concentrations of exhaled, labeled CO2 originating from intravenously administered stable-isotope labeled short-chain fatty acids.
Fecal short-chain fatty acid concentrations by stool samples | Weeks 1, 2, 4, and 5
  Differences and changes in fecal SCFA concentrations in COPD patients and healthy older and young adults.
Body composition by DXA | Weeks 1, 2, 4, and 5
  Differences in muscle mass (kg), fat mass (kg), and bone mineral density (g/cm^2) between COPD patients and healthy older and young adults using DXA.
Bone mineral density by BIA | Weeks 1, 2, 4, and 5
  Differences in muscle mass (kg), fat mass (kg), and extra- and intracellular fluid (L) between COPD patients and healthy older and young adults using BIA.
Handgrip strength dynamometry | Weeks 1, 2, 4, and 5
  Difference and changes in handgrip strength in COPD patients and healthy older and young adults.
6 minute walk test distance | Screening visit
  With this sub-maximal exercise test, aerobic capacity and endurance will be compared between COPD patients and healthy older and young adults. The outcome is the distance covered over a time of 6 minutes.
Skeletal muscle strength of leg | Screening visit
  Difference in muscle strength of leg using kin-com machine between COPD patients and healthy older and young adults.
Micro-respiratory pressure meter measurement | Screening visit
  Difference and changes in maximum inspiratory and expiratory pressure between COPD patients and healthy older and young adults.
C-reactive protein | Weeks 1, 2, 4, and 5
  Differences and changes in the concentration of the inflammatory marker C-reactive protein in COPD patients and healthy older and young adults.
Attention and executive functions measured by Trail Making Test (TMT) | Weeks 1, 2, 4, and 5
  In Part A, the examinee is instructed to connect a set of 25 circles with numbers as quickly as possible while maintaining accuracy. In Part B, the examinee is instructed to connect a set of 25 circles, alternating between numbers and letters, as quickly as possible while maintaining accuracy. Measures attentional resources and is a measure of the frontal lobe "executive" functions of visual search, set-switching and mental flexibility. The total time in seconds will be recorded for each measure.
Attention and executive functions measured by Stroop Color-Word Test (SCWT) | Screening visit
  A word page with words printed in black ink, a color page with blocks printed in color, and a color-word page where the color and the word do not match. The examinee reads the words or names the ink colors as quickly as possible within a time limit. Measures selective attention and inhibitory control. The total time in seconds was reported for each trial.
Gut function as reported by "The Gastrointestinal Symptom Rating Scale" | Weeks 1, 2, 4, and 5
  Self-administered questionnaire regarding gut function and associated symptoms. It is composed of 15 items (7-Point Likert Scale) assessing Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. Scores range from 15 to 105 with a higher score indicating more discomfort.
Physical activity as reported by "Physical Activity Scale for the Elderly" | Weeks 1, 2, 4, and 5
  Self-administered questionnaire is intended for use in an elderly population and focuses on 3 types of activities: leisure time activities, household activities and work-related activities.
State of mood as measured by the Hospital Anxiety and Depression Scale (HADS | Weeks 1, 2, 4, and 5
  A fourteen item self-assessment scale. Seven of the items related to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression.
COPD Assessment Test | Weeks 1, 2, 4, and 5
  Self-administered questionnaire regarding impact of COPD on daily life
3-day diet diary | Completion within the week before study visits of weeks 1, 2, 4, and 5
  The subject is asked to note in detail all the food and drinks consumed during 3 days (2 week days and 1 weekend day) in the week prior to each test day.
Group differences in learning and memory as measured by Digit Span | Weeks 1, 2, 4, and 5
  Recall of numbers in the same order (Digit Forward) and in reverse order (Digit Backward). Measures auditory attention and verbal working memory.
Group differences in overall cognitive abilities as measured by Montreal Cognitive Assessment (MoCA) | Screening visit
  Assesses several cognitive domains and is used for the screening of mild cognitive impairment. Total scores range from 0-30 with lower scores indicating decreased functioning.
Group differences in state of mood as measured by the Profile of Mood State (POMS) | Weeks 1, 2, 4, and 5
  A psychological distress scale to measure mood disturbance in 6 domains - fatigue-inertia, vigor-activity, tension-anxiety, depression-dejection, anger-hostility, and confusion-bewilderment.
Group differences in learning and memory as measured by Controlled Oral Word Association Test (COWAT) | Weeks 1, 2, and 5
  The examinee is required to say as many words as they can think of in one minute that begin with a given letter of the alphabet. The task contains three trials. Measures phonemic verbal fluency. The raw score (total and mean words recorded across the three trials) will be reported.
Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | Weeks 1, 2, 4, and 5
  Quality of life concerns related to fatigue will be assessed only in COPD patients with this questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, Principal Investigator — Texas A&M University - CTRAL
Locations (1):
- Texas A&M University-CTRAL, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kirschner SK, Engelen MP, Haas P, Bischoff SC, Deutz NE. Short-chain fatty acid kinetics and concentrations are higher after inulin supplementation in young and older adults: a randomized trial. Am J Clin Nutr. 2025 Jun;121(6):1224-1235. doi: 10.1016/j.ajcnut.2025.04.018. Epub 2025 Apr 22. PMID 40274191